CLINICAL TRIAL: NCT03464318
Title: Repeatability and Reproducibility of Low-dose Digital Radiographs in the Idiopathic Scoliosis
Brief Title: Low-dose Digital Radiographs in the Idiopathic Scoliosis
Status: Completed | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: RXbd17
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Idiopathic Scoliosis
Keywords: idiopathic scoliosis; radiographs; low dose

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate the intraobserver repeatability and the interobserver reproducibility of low-dose radiographs with a HELIOS DRF (CAT) imaging system in patients with idiopathic scoliosis.

DETAILED DESCRIPTION:
The 80% of scoliosis is idiopathic and begins mostly in adolescence (10-20 years).

The young patients need to undergo several radiographic controls for a correct therapeutic balance. However, the repeated radiation exposures is associated with a greater risk of carcinogenesis even if reduced with a digital imaging technique.

The aim of this study is to evaluate the intraobserver repeatability and the interobserver reproducibility of low-dose radiographs with a HELIOS DRF (CAT) imaging system in patients with idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected or known idiopathic scoliosis
* patients able to maintain orthostasis without medical devices
* patients from 9 to 20 years old

Exclusion Criteria:

* patients with known congenital, syndromic, neurological scoliosis
* patients not able to maintain orthostasis
* obese patients
* low back pain or known tumor pathology
* patients with vertebral arthrodesis
* patients younger than 9 years old, or older than 20 years old

Ages: 9 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: patients with suspected or known idiopathic scoliosis selected at the Rizzoli Orthopaedic Institute
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2018-01-27 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Repeatability and reproducibility | baseline (day 0)
  Repeatability and reproducibility of the Cobb angle measurement

SECONDARY OUTCOMES:
Repeatability and reproducibility | baseline (day 0)
  Repeatability and reproducibility of kyphosis angle, lordosis angle, lumbosacral angle, Nash-Moe rotation index and Risser index measurement
Radiation exposure | baseline (day 0)
  collection of dosimetric data

CONTACTS AND LOCATIONS:
Overall Officials: Milva Battaglia, MD, Principal Investigator — Rizzoli Orthopaedic Institute
Locations (1):
- Rizzoli Orthopaedic Institute, Bologna, Italy